CLINICAL TRIAL: NCT04681131
Title: A Phase 2 Study of BA3011 Alone and in Combination With PD-1 Inhibitor in Adult Patients With Metastatic Non-small Cell Lung Cancer (NSCLC) Who Had Prior Disease Progression on a PD-1/L-1 Inhibitor, EGFR, or ALK Inhibitor.
Brief Title: CAB-AXL-ADC Safety and Efficacy Study in Adults With NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA3011-002
Record Dates: First submitted 2020-12-08; First posted 2020-12-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAB-AXL-ADC (BA3011) (Experimental): CAB-AXL-ADC (BA3011) alone
  Interventions: Biological: CAB-AXL-ADC
- CAB-AXL-ADC (BA3011)+PD-1 inhibitor (Experimental): CAB-AXL-ADC (BA3011) with PD-1 inhibitor
  Interventions: Biological: CAB-AXL-ADC; Biological: PD-1 inhibitor

INTERVENTIONS:
Biological: CAB-AXL-ADC — Conditionally active biologic anti-AXL antibody drug conjugate
  Other Names: BA3011
Biological: PD-1 inhibitor — PD-1 inhibitor
  Arms: CAB-AXL-ADC (BA3011)+PD-1 inhibitor

SUMMARY:
The objective of this study is to assess safety and efficacy of CAB-AXL-ADC in NSCLC

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase 2 study designed to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of BA3011, a conditionally active biologic (CAB) AXL-targeted antibody drug conjugate (CAB-AXL-ADC), alone and in combination with PD-1 inhibitor in patients with metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease.
* Age ≥ 18 years
* Adequate renal function
* Adequate liver function
* Adequate hematological function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least three months.

Exclusion Criteria:

* Patients must not have clinically significant cardiac disease.
* Patients must not have known non-controlled CNS metastasis.
* Patients must not have had prior therapy with a conjugated or unconjugated auristatin derivative/vinca-binding site targeting payload.
* Patients must not have a history of ≥ Grade 3 allergic reactions to mAb therapy as well as known or suspected allergy or intolerance to any agent given during this study.
* Patients must not have had major surgery within 4 weeks before first BA3011
* Patients must not have known human immunodeficiency virus (HIV) infection, active hepatitis B and/or hepatitis C.
* Patients must not be women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) per RECIST v1.1 | Up to 24 months
  Proportion of patients who achieve a confirmed CR or PR according to RECIST v1.1
Incidence of Adverse Events (AEs)or Serious Adverse Events (SAEs) as assessed by CTCAE v4.03/v5 | Up to 24 months
  Measured by frequency and severity of adverse events as assessed by CTCAE v4.03/v5

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 24 months
  Time from the first documented OR until the first documented disease progression or death (due to any cause), whichever occurs first
Progression-free survival (PFS) | Up to 24 months
  Time from the first dose of IP until the first documentation of disease progression or death due to any cause, whichever occurs first.
Best overall response (BOR) | Up to 24 months
  All post-baseline disease assessments that occur prior to the initiation of subsequent anticancer therapy
Disease control rate (DCR) | Up to 24 months
  Proportion of patients with a best overall response of confirmed CR, confirmed PR, or stable disease (SD) ≥ 12 weeks.
Time to response (TTR) | Up to 24 months
  Time from the first dose of investigational product until the first documentation of OR.
Overall survival (OS) | Up to 24 months
  Time from the first dose of BA3021 treatment until death due to any cause.
Percent change from baseline in target lesion sum of diameters | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (60):
- United States (32):
  - City of Hope - Duarte, Duarte, California
  - University of California Irvine Medical Center (UCIMC) - Chao Family Comprehensive Cancer Center, Irvine, California
  - California Research Institute, Los Angeles, California
  - USC Norris, Los Angeles, California
  - Cedars-Sinai, Los Angeles, California
  - University of California, San Diego (UCSD) - Moores Cancer Center, San Diego, California
  - American Institute of Research, Whittier, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Florida Cancer Specialists & Research Institute, Fleming Island, Florida
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Florida Cancer Specialist, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Augusta University - Georgia Cancer Center, Augusta, Georgia
  - Baptist Health Systems, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - Hematology/Oncology Clinic, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Roswell Park, Buffalo, New York
  - NYU Langone Health, New York, New York
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Gabrail Cancer Research Center, Canton, Ohio
  - The Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina- Hollings Cancer Center, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson, Houston, Texas
- Greece (4):
  - Henry Dunant Hospital Center, Athens
  - Metropolitan Hospital Perseus Healthcare Group SA, Piraeus
  - Bioclinic Thessaloniki, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (3):
  - ICON Cancer Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Hong Kong United Oncology Centre, Kowloon
- Italy (5):
  - "IRCCS Osp. Policlinico San Martino Pad Ex microbiologia, stanza 9, 1 piano.", Genoa, Liguria
  - Hospital San Giuseppe Moscati, Avellino
  - European Institute of Oncology (IEO), IRCCS, Milan
  - Santa Maria delle Croci Hospital of Ravenna, Ravenna
  - Integrated University Hospital of Verona, Verona
- Poland (5):
  - MED-Polonia, Sp. z o.o. (LLC), Poznan, Greater Poland Voivodeship
  - Institute of Genetics and Immunology GENIM, Lublin, Lublin Voivodeship
  - Maria Sklodowska-Curie - National Research Institute of Oncology, Warsaw, Masovian Voivodeship
  - Polish Mother's Memorial Hospital-Research Institute, Lodz, Łódź Voivodeship
  - Specialistic Oncologic Hospital NU-MED, Tomaszów Mazowiecki, Łódź Voivodeship
- Spain (6):
  - Hospital Universitario Virgen de Valme, Seville, Andalusia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Catalan Institute of Oncology, Hospital Duran i Reynals, Barcelona, Catalonia
  - University Hospital 12 de Octubre, Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
- Taiwan (5):
  - Kaoshiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided